CLINICAL TRIAL: NCT00922831
Title: Progression of Cognitive, Affective, and Physical Symptoms in Multiple Sclerosis.
Brief Title: Progression of Cognitive and Physical Symptoms in Multiple Sclerosis
Status: Withdrawn | Type: Observational
Why Stopped: Funding not available
Sponsor: MidAmerica Neuroscience Research Foundation at Rowe Neurology Institute (Other)
Collaborators: University of Missouri, Kansas City (Other)
Responsible Party: H. Todd Feaster, PsyD, MidAmerica Neuroscience Institute
Other Study IDs: 080514
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis
Keywords: Cognition, Affective MS symptoms
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to look at multiple sclerosis patients process of awareness, learning, and judging status over a 3 year time period.

DETAILED DESCRIPTION:
Patients with multiple sclerosis (MS) frequently experience cognitive and emotional difficulties. Theses neuropsychiatric symptoms are known to be associated with reduced quality of life. However, little is known about the evolution of MS patients' neuropsychiatric difficulties and how these neuropsychiatric changes may be related to other MS symptoms. The purpose of the present study is to examine MS patients' cognitive and emotional status over time as part of standard neuropsychological evaluations in a private practice setting. MS patients presenting for neuropsychological evaluation at the MidAmerica Neuroscience Institute will be provided with the option of participating in thorough evaluation of their cognitive and affective MS symptoms. They will then be followed clinically and receive re-evaluation over a period of 3 years on a yearly basis. It is hoped that this study will help us obtain a better understanding of the factors associated with worsening cognition in MS. A greater understanding of the factors associated with cognitive and affective decline in MS help could lead to the early identification and treatment of at-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Male/female subjects at least 18 years of age with a diagnosis of Clinically Definite Multiple Sclerosis (CDMS) or Clinically Isolated Syndrome (CIS)as confirmed by a neurologist.
* Subjects must be able to give written informed consent and comply with the study protocol. Subjects must also be able to read, write and understand English.
* Are capable of performing the requirements of the neuropsychological test battery.

Exclusion Criteria:

* As judged by the investigator, any clinically significant, unstable or major concomitant disorder or medications.
* In the opinion of the Investigator should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurology Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hunter T Feaster, PsyD, Principal Investigator — MidAmerica Neuroscience Research Foundation at Rowe Neurology Institute; Jared Bruce, PhD, Principal Investigator — University of Missouri, Kansas City